CLINICAL TRIAL: NCT01205841
Title: A Prospective Study Comparing Different Clinical Decision Rules in Adult and Pediatric Ankle Trauma
Acronym: LEFO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Dimitri Vandoninck MD, Emergency Department of the University Hospitals, Catholic University Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S52510
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Ankle Injuries
Keywords: Ottawa Ankle and Foot Rules; Buffalo Rule; Bernese Ankle Rules; Low Risk Exam; Malleolar Zone Algorithm; Clinical decision rule; Ankle injury; Ankle sprain; Inversion trauma
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adults (Experimental): Patients from 16 years of age onwards
  Interventions: Procedure: Ottawa Ankle and Foot Rules; Procedure: Buffalo Rule; Procedure: Ottawa Ankle and Foot Rules + application of a tuning fork to the distal fibula and tibia; Procedure: Thompson Test; Procedure: Palpation of the fibula; Procedure: Bernese Ankle Rules
- Children (Experimental): Patients aged 5 to 15 years
  Interventions: Procedure: Ottawa Ankle and Foot Rules; Procedure: Buffalo Rule; Procedure: Ottawa Ankle and Foot Rules + application of a tuning fork to the distal fibula and tibia; Procedure: Thompson Test; Procedure: Palpation of the fibula; Procedure: Ottawa Ankle and Foot Rules + palpation of the cuboid bone; Procedure: Ottawa Ankle and Foot Rules + palpation over the deltoid ligament; Procedure: Malleolar Zone Algorithm; Procedure: Low Risk Exam; Procedure: Bernese Ankle Rules; Procedure: Ottawa Ankle and Foot Rules + swelling of the distal fibula

INTERVENTIONS:
Procedure: Ottawa Ankle and Foot Rules — As previously published
Procedure: Buffalo Rule — As previously published
Procedure: Ottawa Ankle and Foot Rules + application of a tuning fork to the distal fibula and tibia — As previously published
Procedure: Thompson Test — As previously published
Procedure: Palpation of the fibula — Palpation of the fibula over its entire length.
Procedure: Ottawa Ankle and Foot Rules + palpation of the cuboid bone — As previously published
  Arms: Children
Procedure: Ottawa Ankle and Foot Rules + palpation over the deltoid ligament — As previously published
  Arms: Children
Procedure: Malleolar Zone Algorithm — As previously published
  Arms: Children
Procedure: Low Risk Exam — As previously published
  Arms: Children
Procedure: Bernese Ankle Rules — As previously published
Procedure: Ottawa Ankle and Foot Rules + swelling of the distal fibula — As previously published
  Arms: Children

SUMMARY:
Comparison of the reliability of different examination techniques to detect fractures in patients with ankle trauma.

DETAILED DESCRIPTION:
Patients with ankle trauma frequently present in the emergency department. In many institutions radiographies of the ankle and foot are obtained in most of these patients, although significant fractures occur only in 15%. Therefore clinical decision rules were developed to clinically rule out significant ankle fractures, thereby reducing the number of radiographies resulting in significant time and cost savings.

Up until now the Ottawa Ankle and Foot Rules are the only clinical decision rules for ankle trauma that are widely accepted. They have a high sensitivity for the detection of fractures but a relatively low specificity. This led to the development of alternative clinical decision rules claiming equally high sensitivity but improved specificity. These alternatives have mostly not been replicated nor have they been directly compared.

This is what the researchers want to do in this study: compare different clinical decision rules regarding sensitivity and specificity. Radiographies of ankle and foot made for every patient are used as the gold standard for the detection of fractures.

Different clinical decision rules will be compared in a pediatric (5-15 years) and an adult population (from 16 years onwards). The researchers consider a clinical decision rule acceptable of it has a sensitivity of at least 95% and a specificity of at least 25%.

ELIGIBILITY:
Inclusion Criteria:

* Pain due to blunt trauma to the ankle
* Must be at least 5 years old

Exclusion Criteria:

* Skin defects in the injured area
* Time of trauma > 72 hours before presentation
* Multiple significant injuries making clinical examination impossible
* Clinically obvious fracture
* Re-evaluation
* Referred with radiography
* Result of radiography already known to investigator
* Glasgow Coma Scale < 15

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for detection of significant fractures | At the first visit to the emergency department
  * In the adult population: fractures of the ankle, midfoot or fibula with a fragment measuring > 3mm detected by radiography
  * In the pediatric population: fractures of the ankle, midfoot or fibula with a fragment measuring > 3mm detected by radiography. Salter-Harris I and II are not considered to be significant fractures. Due to considerable controversy in the literature sensitivity and specificity of the clinical decision rules will be calculated separately for different definitions of significant fractures.
Specificity for detection of significant fractures | At the first visit to the emergency department
  * In the adult population: fractures of the ankle, midfoot or fibula with a fragment measuring > 3mm detected by radiography
  * In the pediatric population: fractures of the ankle, midfoot or fibula with a fragment measuring > 3mm detected by radiography. Salter-Harris I and II are not considered to be significant fractures. Due to considerable controversy in the literature sensitivity and specificity of the clinical decision rules will be calculated separately for different definitions of significant fractures.

SECONDARY OUTCOMES:
Prevalence of proximal fibula fractures in ankle trauma | At the first visit to the emergency department
  The prevalence of proximal fibula fractures in ankle trauma has, to the best of our knowledge, not yet been quantified.
Prevalence of gastrocnemius tendon rupture in ankle trauma | At the first visit to the emergency department
  The prevalence of gastrocnemius tendon rupture in ankle trauma has, to the best of our knowledge, not yet been quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Vandoninck, MD, Principal Investigator — Emergency Department of the University Hospitals, Catholic University Leuven; Marc Sabbe, MD, PhD, Study Director — Emergency Department of the University Hospitals, Catholic University Leuven
Locations (1):
- Emergency Department of the University Hospitals, Catholic University Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Eggli S, Sclabas GM, Eggli S, Zimmermann H, Exadaktylos AK. The Bernese ankle rules: a fast, reliable test after low-energy, supination-type malleolar and midfoot trauma. J Trauma. 2005 Nov;59(5):1268-71. doi: 10.1097/01.ta.0000196436.95569.a3. PMID 16385314
- [Background] Dissmann PD, Han KH. The tuning fork test--a useful tool for improving specificity in "Ottawa positive" patients after ankle inversion injury. Emerg Med J. 2006 Oct;23(10):788-90. doi: 10.1136/emj.2006.035519. PMID 16988308
- [Background] Leddy JJ, Kesari A, Smolinski RJ. Implementation of the Ottawa ankle rule in a university sports medicine center. Med Sci Sports Exerc. 2002 Jan;34(1):57-62. doi: 10.1097/00005768-200201000-00010. PMID 11782648
- [Background] Stiell IG, Greenberg GH, McKnight RD, Nair RC, McDowell I, Worthington JR. A study to develop clinical decision rules for the use of radiography in acute ankle injuries. Ann Emerg Med. 1992 Apr;21(4):384-90. doi: 10.1016/s0196-0644(05)82656-3. PMID 1554175
- [Background] Dayan PS, Vitale M, Langsam DJ, Ruzal-Shapiro C, Novick MK, Kuppermann N, Miller SZ. Derivation of clinical prediction rules to identify children with fractures after twisting injuries of the ankle. Acad Emerg Med. 2004 Jul;11(7):736-43. doi: 10.1197/j.aem.2004.02.517. PMID 15231460
- [Background] Boutis K, Komar L, Jaramillo D, Babyn P, Alman B, Snyder B, Mandl KD, Schuh S. Sensitivity of a clinical examination to predict need for radiography in children with ankle injuries: a prospective study. Lancet. 2001 Dec 22-29;358(9299):2118-21. doi: 10.1016/S0140-6736(01)07218-X. PMID 11784626
- [Background] Clark KD, Tanner S. Evaluation of the Ottawa ankle rules in children. Pediatr Emerg Care. 2003 Apr;19(2):73-8. doi: 10.1097/00006565-200304000-00003. PMID 12698029